CLINICAL TRIAL: NCT04530591
Title: A Proof of Concept, Randomized, Single Center Study on Frameworks for Wearable Devices to Sense and Respond to Opioid Overdoses
Brief Title: User Acceptability of a Device-Based Opioid Overdose Intervention
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 834304
Record Dates: First submitted 2020-08-24; First posted 2020-08-28 (Actual); Results first posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Opioid Overdose; Opioid-use Disorder; Substance Use Disorders
Keywords: Naloxone Delivery; Survey
MeSH Terms: conditions — Opiate Overdose; Opioid-Related Disorders; Substance-Related Disorders | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient Participants: This group of participants will complete a survey about their opioid use history and their preferences for a device-based intervention. They will then participate in a semi-structured interview to provide feedback on non-functional, "looks-like" prototypes of such a device.
  Interventions: Other: Survey; Other: Interview

INTERVENTIONS:
Other: Survey — Participants will complete a survey about their opioid use history, its impact on their lives, their current strategies for preventing or reversing opioid overdoses, and their preferences for a device-based intervention.
Other: Interview — Participants will participate in a semi-structured interview, during which they will provide feedback on non-functional, "looks-like" prototypes of a naloxone delivery device.

SUMMARY:
This pilot study evaluates the needs of opioid users for a device-based intervention for opioid overdoses. The results of this one-time short questionnaire will inform development of a novel naloxone delivery device.

DETAILED DESCRIPTION:
All opioid overdose related deaths can be prevented with the timely delivery of Naloxone. This study is a one-time, preliminary survey of participants with opioid use disorder to assess the need for, and community attitudes towards, a wearable device capable of autonomously detecting and responding to an opioid overdose. The results of this survey will be used to guide ongoing development of a de novo device. This study will be conducted over a 3 month period and survey participants from the Kensington Neighborhood in North Philadelphia.

ELIGIBILITY:
Inclusion Criteria:

* Have used opioids for more than 3 months or will be having surgery where opioids will be administered

  * Able to provide informed consent
  * Moderate to severe chronic pain treated with opioids or recreational use

Exclusion Criteria:

* Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is non-pregnant individuals over the age of 21 with opioid use disorder.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Brenner, MD/PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Prevention Point Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kanter K, Gallagher R, Eweje F, Lee A, Gordon D, Landy S, Gasior J, Soto-Calderon H, Cronholm PF, Cocchiaro B, Weimer J, Roth A, Lankenau S, Brenner J. Willingness to use a wearable device capable of detecting and reversing overdose among people who use opioids in Philadelphia. Harm Reduct J. 2021 Jul 23;18(1):75. doi: 10.1186/s12954-021-00522-3. PMID 34301246

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patient Participants
Started | 97
Completed | 97
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patient Participants
Number analyzed (Participants) | 97
Age, Continuous [Mean (Inter-Quartile Range); unit: Years] | 41 [37 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23
  Not Hispanic or Latino | 74
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 30
  White | 46
  More than one race | 0
  Unknown or Not Reported | 20
Housing Status [Count of Participants; unit: Participants]
  Homeless | 31
  House | 7
  Apartment | 8
  Shelter | 36
  Unknown | 15
Started After Injury/Surgery [Count of Participants; unit: Participants]
  Yes | 46
  No | 51
Duration of Opioid Use [Mean (Inter-Quartile Range); unit: years] | 12 [8 to 20]
Opioid Use Frequency (Days per Week) [Count of Participants; unit: Participants]
  1 | 0
  2-3 | 9
  4-6 | 7
  7 | 80
  Unknown | 1
Opioid Use Frequency (Uses per Day) [Count of Participants; unit: Participants]
  1 | 1
  2-3 | 21
  4-6 | 46
  7+ | 27
  Unknown | 2
Been to an Inpatient Rehab [Count of Participants; unit: Participants]
  Yes | 79
  No | 18
Used MOUD [Count of Participants; unit: Participants]
  Yes | 84
  No | 13
Perceived likelihood of bystander intervention in the event of an overdose [Count of Participants; unit: Participants]
  Likely | 53
  Unlikely | 44
Friends/Family Who have Overdosed [Count of Participants; unit: Participants]
  Yes | 77
  No | 20
Friends/Family Who have had Overdose Complications [Count of Participants; unit: Participants]
  Yes | 56
  No | 41
Friends/Family Who have Died from Overdose [Count of Participants; unit: Participants]
  Yes | 75
  No | 22
Has Overdosed [Count of Participants; unit: Participants]
  Yes | 69
  No | 28
Number of Prior Overdoses [Mean (Inter-Quartile Range); unit: Incidents] | 3 [2 to 7]

OUTCOME MEASURES:

1. Primary Outcome: Community Need for a Device-based Opioid Overdose Intervention
Description: We aim to characterize the degree of need for a device-based opioid overdose intervention. These were extracted from the participant survey questions as well as from the words, phrases, and sentences used by participants during the interview.
Time Frame: Day 1
Population: Some participants did not answer all the questions or selected more than one answer
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Participants
Number analyzed (Participants) | 91
Participants
  Likely | 69
  Unlikely | 22

2. Secondary Outcome: Functional and Aesthetic Preferences for Device-based Opioid Overdose Intervention
Description: We aim to characterize the functional and aesthetic preferences of the participant population for a device-based opioid overdose intervention. These were extracted from the participant survey questions as well as from the words, phrases, and sentences used by participants during the interview.
Time Frame: Day 1
Population: Some participants did not answer all the questions or selected more than one answer
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Participants
Number analyzed (Participants) | 97
Participants
  Likely to use a device that senses an overdose: number analyzed (Participants) | 96
  Likely to use a device that senses an overdose: Likely | 70
  Likely to use a device that senses an overdose: Unlikely | 26
  Likely to use a device that indicates the wearer is at risk of an overdose: number analyzed (Participants) | 95
  Likely to use a device that indicates the wearer is at risk of an overdose: Likely | 66
  Likely to use a device that indicates the wearer is at risk of an overdose: Unlikely | 29
  Likely to use a device that straps naloxone to the body for a bystander to administer: number analyzed (Participants) | 96
  Likely to use a device that straps naloxone to the body for a bystander to administer: Likely | 52
  Likely to use a device that straps naloxone to the body for a bystander to administer: Unlikely | 44
  Likely to use a device that senses an overdose and administers naloxone if needed: number analyzed (Participants) | 96
  Likely to use a device that senses an overdose and administers naloxone if needed: Likely | 64
  Likely to use a device that senses an overdose and administers naloxone if needed: Unlikely | 32
  Likely to use a device that alerts medical first responders if needed: number analyzed (Participants) | 96
  Likely to use a device that alerts medical first responders if needed: Likely | 68
  Likely to use a device that alerts medical first responders if needed: Unlikely | 28
  Likely to use a device that alerts bystanders if needed: number analyzed (Participants) | 95
  Likely to use a device that alerts bystanders if needed: Likely | 60
  Likely to use a device that alerts bystanders if needed: Unlikely | 35
  Likely to use a device that monitors vital signs: number analyzed (Participants) | 95
  Likely to use a device that monitors vital signs: Likely | 73
  Likely to use a device that monitors vital signs: Unlikely | 22
  For a device that sense overdose - likely to wear a necklace: number analyzed (Participants) | 94
  For a device that sense overdose - likely to wear a necklace: Likely | 48
  For a device that sense overdose - likely to wear a necklace: Unlikely | 46
  For a device that sense overdose - likely to wear a canula: number analyzed (Participants) | 96
  For a device that sense overdose - likely to wear a canula: Likely | 12
  For a device that sense overdose - likely to wear a canula: Unlikely | 84
  For a device that sense overdose - likely to wear a skin-patch on chest: number analyzed (Participants) | 96
  For a device that sense overdose - likely to wear a skin-patch on chest: Likely | 42
  For a device that sense overdose - likely to wear a skin-patch on chest: Unlikely | 54
  For a device that sense overdose - likely to wear a skin-patch on upper arm: number analyzed (Participants) | 96
  For a device that sense overdose - likely to wear a skin-patch on upper arm: Likely | 53
  For a device that sense overdose - likely to wear a skin-patch on upper arm: Unlikely | 43
  For a device that sense overdose - likely to wear a watch-appearing bracelet: number analyzed (Participants) | 94
  For a device that sense overdose - likely to wear a watch-appearing bracelet: Likely | 72
  For a device that sense overdose - likely to wear a watch-appearing bracelet: Unlikely | 22
  For a device that sense overdose - likely to wear a wrist bracelet: number analyzed (Participants) | 95
  For a device that sense overdose - likely to wear a wrist bracelet: Likely | 69
  For a device that sense overdose - likely to wear a wrist bracelet: Unlikely | 26
  For a device that sense overdose - likely to wear a shoulder strap: number analyzed (Participants) | 51
  For a device that sense overdose - likely to wear a shoulder strap: Likely | 21
  For a device that sense overdose - likely to wear a shoulder strap: Unlikely | 30
  For a device that sense overdose - likely to wear a thigh strap: number analyzed (Participants) | 48
  For a device that sense overdose - likely to wear a thigh strap: Likely | 15
  For a device that sense overdose - likely to wear a thigh strap: Unlikely | 33
  For a device that sense overdose - likely to wear a chest strap: number analyzed (Participants) | 94
  For a device that sense overdose - likely to wear a chest strap: Likely | 22
  For a device that sense overdose - likely to wear a chest strap: Unlikely | 72
  For a device that sense overdose - likely to wear glasses: number analyzed (Participants) | 94
  For a device that sense overdose - likely to wear glasses: Likely | 24
  For a device that sense overdose - likely to wear glasses: Unlikely | 70
  For a device that sense overdose - likely to wear a knee brace: number analyzed (Participants) | 48
  For a device that sense overdose - likely to wear a knee brace: Likely | 16
  For a device that sense overdose - likely to wear a knee brace: Unlikely | 32
  For a device that sense overdose - likely to wear an ankle strap: number analyzed (Participants) | 96
  For a device that sense overdose - likely to wear an ankle strap: Likely | 44
  For a device that sense overdose - likely to wear an ankle strap: Unlikely | 52

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at the time of survey administration (1 hour).
Description: Participants were asked to complete a survey and participate in an interview. There is no risk for mortality or serious adverse events from these activities.
Arm/Group | Patient Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/97

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/91/NCT04530591/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/91/NCT04530591/ICF_001.pdf